CLINICAL TRIAL: NCT02659332
Title: Diode Laser Treatment of Pta Low Grade Bladder Tumors in the Outpatient Department
Brief Title: Laser Treatment of Bladder Tumors in the Outpatient Department
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Gregers G Hermann (Other)
Responsible Party: Sponsor-Investigator, Gregers G Hermann, MD, DM Sc., Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URU05
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Bladder Tumors
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TURBT (Experimental): Diode laser (400μm fiber, 6-12W, laser pulse 1ms and intervals of1ms)
  Interventions: Device: TURBT

INTERVENTIONS:
Device: TURBT — Diode laser (400μm fiber, 6-12W, laser pulse 1ms and intervals of 1 ms)

SUMMARY:
* Primary Objective: To show that small pTa bladder tumors can be removed with diode laser in an outpatient department.
* Secondary Objective: To evaluate the patients' symptoms during and after the laser TURBT.
* Tertiary Objective: To evaluate the rate of remnant tumor tissue one month after the laser TURBT.

DETAILED DESCRIPTION:
The patients will have a PDD guided flexible cystoscopy performed and the bladder tumor will be removed by a diode laser (400μm fiber, 6-12W, laser pulse 1ms and intervals of1ms).The treatment will take place in the OPD in awaken patients. One hour prior to the treatment the patient will have Hexvix® (photodynamic substance) and Lidocaine 20 ml (pain treatment) installed in the bladder. Simultaneous pain treatment will be oral Paracetamol 1 g and Ibuprofen 600 mg. Biopsy from the tumor will be taken to confirm the histological diagnosis.

Immediately after the procedure the pain assessed by the VAS score will be recorded and the patients are given a QOL questionnaire (EORTC QLQ-BLS24) and a stamped envelope and are asked to return it one week later. The patients will be telephoned after 5 days to remind on the questionnaire and to ash, whether they has had a urinary infection after the procedure.

One month after the laser TURBT a flexible PPD and SPIES guided cystoscopy is performed in the OPD to evaluate the laser efficacy. To confirm that all tumour tissue has been removed a biopsy will be taken from the previous tumor place. The biopsy will be send to the pathologist according to the normal procedure for biopsies. Visual presentation of the laser treated area will be visualized using PDD and SPIES.

ELIGIBILITY:
Inclusion Criteria:

* Recurrence of pTa low grade urothelial bladder tumor
* Tumor < 1.5 cm
* < 6 tumors

Exclusion Criteria:

* Patients with porphyria
* Known hypersensitivity to Hexvix® or porfhyrins
* Use of any anticoagulantia
* Macroscopic hematuria
* Pregnant or breast feeding women
* Expected poor compliance
* Patients < 18 years
* Patients who do not read or understand Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-03 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Complete Removal by One Laser Treatment (Proportions of patients where the bladder tumors are completely removed by one laser) | one month
  Proportions of patients where the bladder tumors are completely removed by one laser treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gregers G Hermann, MD, DMSc, Principal Investigator — Bispebjerg and Frederiksberg Hospital
Locations (1):
- Department of Urology, Bispebjerg and Frederiksberg Hospital, Frederiksberg, Copenhagen, Denmark

REFERENCES:
- [Background] Ferlay J, Steliarova-Foucher E, Lortet-Tieulent J, Rosso S, Coebergh JW, Comber H, Forman D, Bray F. Cancer incidence and mortality patterns in Europe: estimates for 40 countries in 2012. Eur J Cancer. 2013 Apr;49(6):1374-403. doi: 10.1016/j.ejca.2012.12.027. Epub 2013 Feb 26. PMID 23485231
- [Background] Sangar VK, Ragavan N, Matanhelia SS, Watson MW, Blades RA. The economic consequences of prostate and bladder cancer in the UK. BJU Int. 2005 Jan;95(1):59-63. doi: 10.1111/j.1464-410X.2005.05249.x. PMID 15638895
- [Background] van Rhijn BW, Burger M, Lotan Y, Solsona E, Stief CG, Sylvester RJ, Witjes JA, Zlotta AR. Recurrence and progression of disease in non-muscle-invasive bladder cancer: from epidemiology to treatment strategy. Eur Urol. 2009 Sep;56(3):430-42. doi: 10.1016/j.eururo.2009.06.028. Epub 2009 Jun 26. PMID 19576682
- [Background] James AC, Gore JL. The costs of non-muscle invasive bladder cancer. Urol Clin North Am. 2013 May;40(2):261-9. doi: 10.1016/j.ucl.2013.01.004. Epub 2013 Feb 13. PMID 23540783
- [Background] Hofstetter A, Frank F, Keiditsch E, Bowering R. Endoscopic Neodymium-YAG laser application for destroying bladder tumors. Eur Urol. 1981;7(5):278-82. doi: 10.1159/000473240. PMID 6894732
- [Background] Davenport K, Keeley FX Jr, Timoney AG. Audit of safety, efficacy, and cost-effectiveness of local anaesthetic cystodiathermy. Ann R Coll Surg Engl. 2010 Nov;92(8):706-9. doi: 10.1308/003588410X12699663904835. Epub 2010 Jul 2. PMID 20615299
- [Background] Syed HA, Talbot N, Abbas A, MacDonald D, Jones R, Marr TJ, Rukin NJ. Flexible cystoscopy and Holmium:Yttrium aluminum garnet laser ablation for recurrent nonmuscle invasive bladder carcinoma under local anesthesia. J Endourol. 2013 Jul;27(7):886-91. doi: 10.1089/end.2012.0696. Epub 2013 Jun 22. PMID 23537221
- [Background] Wong KA, Zisengwe G, Athanasiou T, O'Brien T, Thomas K. Outpatient laser ablation of non-muscle-invasive bladder cancer: is it safe, tolerable and cost-effective? BJU Int. 2013 Sep;112(5):561-7. doi: 10.1111/bju.12216. Epub 2013 Jul 2. PMID 23819486
- [Background] Hermann GG, Mogensen K, Toft BG, Glenthoj A, Pedersen HM. Outpatient diagnostic of bladder tumours in flexible cystoscopes: evaluation of fluorescence-guided flexible cystoscopy and bladder biopsies. Scand J Urol Nephrol. 2012 Feb;46(1):31-6. doi: 10.3109/00365599.2011.637954. Epub 2011 Dec 12. PMID 22150596
- [Background] Turrentine FE, Wang H, Simpson VB, Jones RS. Surgical risk factors, morbidity, and mortality in elderly patients. J Am Coll Surg. 2006 Dec;203(6):865-77. doi: 10.1016/j.jamcollsurg.2006.08.026. PMID 17116555